CLINICAL TRIAL: NCT06833762
Title: Determining Clinical and Cardiopulmonary Exercise Testing Parameters That Predict Improvement in Functional Capacity and Complications After Transcatheter Aortic Valve Implantation
Brief Title: Clinical and CPET Parameters That Predict Improvement in Functional Capacity After TAVI
Status: Recruiting | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: TAVI-CPET
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-10

CONDITIONS: Aortic Stenosis Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Determining Clinical and Cardiopulmonary exercise testing Parameters that may predict Improvement in Capacity After Transcatheter Aortic Valve Implantation

DETAILED DESCRIPTION:
Transcatheter Aortic Valve Implantation (TAVI) has emerged as a less invasive alternative to surgical aortic valve replacement, especially for high-risk patients. However, existing research on functional outcomes after TAVI has yielded mixed results. To our knowledge, the potential functional benefit of TAVI has not been well explored using cardiopulmonary exercise testing (CPET). The present study aims to 1) characterize the mid-term exercise tolerance response to TAVI, and 2) determine the clinical (symptoms, frailty, quality of life, etc.) and functional factors (parameters derived from CPET) that determine the magnitude of this response. A positive functional response to TAVI will be considered as an increase in VO2 max > 2.5ml/kg/min or >10% of its baseline value one month post-TAVI. The exercise test will be conducted by a physiotherapist and supervised by a physician using a standard incremental cardiopulmonary exercise testing on cycle ergometer (Ergoline 900, Ergoline, Bitz, Germany (CE-0123) and Ergocard Professional, Medisoft, Sorinnes, Belgium (CE-1434)). To this end, 161 patients with severe aortic stenosis scheduled for TAVI will be included in 3 expert centres. They will be evaluated clinically and functionally (incremental CPET) in the 2 weeks prior to the procedure and 4-6 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* All those patients ≥ 18 years of age with severe aortic stenosis approved for transfemoral TAVI.

Both sexes, male and female will be included in the study.

Exclusion Criteria:

Very severe aortic stenosis, defined as a valve area of ≤0.6 cm2

, mean gradient ≥60 mmHg or Vmax >5 m/s

* Previous syncope
* Proven exercise-induced arrhythmias
* Previously known dynamic left ventricular outflow tract (LVOT) obstruction, defined as LVOT gradient of ≥ 30 mmHg by echocardiography
* Concomitant coronary artery disease pending percutaneous coronary intervention
* Inability to consent
* Physical limitation to perform an exercise test
* Non-elective procedure
* Valve-in-valve procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Study Population: Patients 18 years of age or older, with severe, non-critical, aortic stenosis who are scheduled for transfemoral TAVI will participate in the study
Sampling Method: Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Delta VO2 max and Delta VO2 at anaerobic threshold | CPET performed 2 weeks before TAVI and 4-6 weeks after
  Change in CPET parameters after Transcatheter Aortic valve implantation (TAVI): VO2 max, VO2 at anaerobic threshold
Clinical and functional pre-TAVI factors that predict improvement in functional capacity after TAVI | CPET performed 2 weeks before TAVI and 4-6 weeks after
  To identify clinical and functional pre-TAVI factors that predict improvement in functional capacity after TAVI (i.e., VO2 max increase > 2.5 ml/kg/min or >10% increase in VO2 max).
  ml/kg/min or >10% increase in VO2 max).

SECONDARY OUTCOMES:
Clinical predictors of improvement in quality of life | 2 weeks before TAVI and 4-6 weeks after
  To identify clinical, echocardiographic and functional pre-TAVI variables that predict improvement in quality of life
pre-TAVI CPET parameters that predict in-hospital complications. | CPET performed 2 weeks before TAVI and 4-6 weeks after
  Correlation between pre-TAVI CPET parameters and in-hospital complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain